CLINICAL TRIAL: NCT04575558
Title: A Randomized, Multi-institutional, Phase 2 Study of Hydroxichloroquine Plus Azithromycin for High Risk SARS-CoV-2 Positive Patients (COVID-19)
Brief Title: HOPE: A Trial of Hydroxichloroquine Plus Azithromycin in High Risk COVID-19
Acronym: HOPE_BRAZIL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to lack of study centers interested in participating.
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Oncoclínicas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LACOG 0220
Record Dates: First submitted 2020-05-18; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Sars-CoV2
MeSH Terms: interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine + Azithromycin (Experimental): Hydroxychloroquine 400mg PO BID 2 times a day + Azithromycin 500mg PO QD, both for 7 days
  Interventions: Drug: Hydroxychloroquine and Azithromycin
- Hydroxychloroquine + Placebo tablets (Placebo Comparator): Hydroxychloroquine 400mg PO BID 2 times a day + Placebo, both for 7 days
  Interventions: Drug: Hydroxychloroquine and Azithromycin

INTERVENTIONS:
Drug: Hydroxychloroquine and Azithromycin — Hydroxychloroquine 400mg PO BID 2 times a day + Azithromycin 500mg PO QD
  Other Names: Reuquinol + Zitromax

SUMMARY:
Multicenter, double blind, randomized clinical trial for high-risk patients over 18 years of age, symptomatic for COVID-19 infection, without any severity criteria

DETAILED DESCRIPTION:
COVID-19 is a respiratory disease caused by a new coronavirus (SARS-CoV2) and with substantial morbidity and mortality. Among different populations at risk, cancer patients stand out. These patients undergo immunosuppressive treatments with chemotherapy and radiotherapy and more often require hospital visit for treatment and monitoring.

Several strategies have been investigated to deal with this situation. Antiretrovirals, anti-inflammatories, antibiotics, anti-IL6, immune response modulating agents, among others, including combinations. Most of these experiences have focused on patients with severe hospitalized conditions

As of March 28, approximately 630,000 confirmed cases have been recorded, including 24,282 serious cases and 28,963 deaths worldwide. In Brazil, after one month since the first case, there are 3417 infected and 92 deaths. All states registered cases of the disease, and nine have deaths: Amazonas, Ceará, Pernambuco, Rio de Janeiro, Goiás, Paraná, Santa Catarina, Rio Gran de do Sul and São Paulo. Cases have progressed and currently there is no specific antiviral therapy for coronavirus infections. A few intervention studies have been conducted as most strains of human coronavirus cause self-limiting diseases and requires only supportive care. After the severe acute respiratory syndrome (SARS), the coronavirus was identified in 2002 and caused a major global outbreak, there was a growing interest in the development of specific therapeutic agents. Therefore, since the SARS outbreak, new therapeutic agents targeting viral entry, proteins, proteases, polymerases and methyltransferases have been tested. Nevertheless, none of them have been shown to be effective in clinical trials. Recent publications have drawn attention to the possible benefit of drugs such as chloroquine, hydroxychloroquine associated or not with azithromycin, which have been used in the treatment of patients infected with SARS- CoV.

Using the combination of hydroxychloroquine and azithromycin, French patients confirmed with Covid-19 were included in a single arm protocol between early March and March 16th, receiving 600mg of hydroxychloroquine daily. Nasal swab viral load was tested daily in a hospital setting. Azithromycin was added to the treatment based on the clinical presentation. Control patients included patients from another center and those who refused the protocol. Day End point was presence or absence of virus on day 6 post-inclusion. There were six asymptomatic patients, twnty two with upper respiratory tract infection and eight had symptoms of lower respiratory tract infection. Twenty cases were treated in this study and showed a significant reduction in viral transport at post-day 6 of inclusion compared to controls, and mean transport duration much shorter than that reported in untreated patients in the literature. Despite the small sample size, research shows that treatment with hydroxychloroquine is associated with a significantly reduction / disappearance of viral load in patients with COVID-19, and its effect seems to be reinforced by azithromycin.

Hydroxychloroquine alone or in combination with azithromycin has been increasingly studied and used in the treatment of respiratory disease induced by COVID-19. In March 2020, the Food and Drug Administration (FDA) interim approved the use of the combination of hydroxychloroquine and azithromycin for clinical use in patients with severe respiratory syndrome associated with coronavirus. There are dozens of studies in progress evaluating this therapeutic alternative in different regions of the world. The World Health Organization (WHO) has just launched a global clinical trial evaluating the four treatments considered promising, including hydroxychloroquine. In Brazil, a consortium of clinical research is underway that is conducting three randomized clinical trials with treatments with hydroxychloroquine, azithromycin and corticosteroids. Considering that these medications have been studied in different institutions and regions and in different contexts, it is important to know the role that these medications can play in the prevention or treatment of COVID-19 in a population of cancer patients undergoing cancer treatments such as chemotherapy and immunotherapy.This clinical trial was designed to evaluate the therapeutic effect of the combination of hydroxychloroquine and azithromycin on non-critical adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and by 1 of the following criteria:

  1. Cancer diagnosis and systemic antineoplastic treatment (chemotherapy or hormone therapy or immunotherapy or small molecule therapy), or having received the last dose within 90 days from randomization, or
  2. Antineoplastic treatment with radiotherapy or had received the last fraction within 90 days from randomization, or
  3. Undergone surgery for cancer treatment within 90 days from randomization, or
  4. Need for continuous treatment for chronic disease. asthma, COPD, pulmonary fibrosis, pulmonary hypertension, smoking, systemic arterial hypertension, ischemic heart disease, hypertensive heart disease, symptomatic valve heart disease, cardiac arrhythmia, chronic renal failure, stroke, diabetes, autoimmune or other disease at the discretion of the investigator.
* Confirmed diagnosis of SARS-CoV-2 infection;
* Symptoms of SARS-Cov-2 (COVID-19) infection but without showing signs / symptoms of severity;
* Respiratory rate <24ipm;
* HR <130 bpm (in the absence of fever);
* Oxygen saturation > 90%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Clinical deterioration rate | 37 days
  Clinical deterioration throughout treatment

SECONDARY OUTCOMES:
Mortality and cause of death | 60 days
  Evaluate the mortality and cause of death, at the end of treatment, at 28 days and 60 days from the start of treatment
Incidence and type of Adverse Events (EAs) | 37 days
Incidence and type of Serious Adverse Events (SAE) | 37 days
Discontinuation rate or temporary suspension of treatment | 37 days
Descriptive radiologic changes on chest CT scans | 37 days

CONTACTS AND LOCATIONS:
Locations (7):
- Brazil (7):
  - Núcleo de Oncologia da Bahia - NOB, Salvador, Estado de Bahia
  - Oncoclínicas BH, Belo Horizonte, Minas Gerais
  - Centro Oncológico do Triângulo - COT, Uberlândia, Minas Gerais
  - Multihemo, Recife, Pernambuco
  - Oncoclinicas RJ, Rio de Janeiro, Rio de Janeiro
  - Centro de Pesquisa em Oncologia PUCRS, Porto Alegre, Rio Grande do Sul
  - Centro Paulista de Oncologia, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No